CLINICAL TRIAL: NCT04082481
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Rising Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAK-988 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of TAK-988 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study stopped early, before enrolling its first participant.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: TAK-988-1001; U1111-1238-5474 (Registry Identifier: WHO)
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TAK-988: Part A (Experimental): TAK-988 tablet or TAK-988 placebo-matching tablet, orally, once on Day 1 to healthy non-Japanese participants. Sentinel dosing will be done in the first 2 cohorts of Part A (Cohorts A1 and A2 [fasted and fed dosing conditions]). Dose escalation in Cohorts A2 to A6 will be based on emerging safety/tolerability, PK, and PD data from previous cohorts.
  Interventions: Drug: TAK-988; Drug: TAK-988 Placebo
- TAK-988: Part B (Experimental): TAK-988 tablet or TAK-988 placebo-matching tablet, orally, twice daily (6-hour interval) from Day 1 to Day 14 to healthy non-Japanese participants. Dose escalation will be based on review of the emerging safety/tolerability, PK, and PD data from previous cohorts and Part A.
  Interventions: Drug: TAK-988; Drug: TAK-988 Placebo
- TAK-988: Part C (Experimental): TAK-988 tablet or TAK-988 placebo-matching tablet, orally, twice daily (6-hour interval) from Day 1 to Day 7 to healthy non-Japanese participants. Dose will be determined based on previous multiple-rising dose (MRD) cohorts.
  Interventions: Drug: TAK-988; Drug: TAK-988 Placebo
- TAK-988: Part D (Experimental): TAK-988 tablet or TAK-988 placebo-matching tablet, orally, twice daily (6-hour interval) from Day 1 to Day 14 to HE non-Japanese participants. Dose will be determined based on previous MRD cohorts.
  Interventions: Drug: TAK-988; Drug: TAK-988 Placebo
- TAK-988: Part E (Experimental): TAK-988 tablet or TAK-988 placebo-matching tablet, orally, once on Day 1, followed by a washout period of 2 days and twice daily (6- hour interval) on Day 3 and continue to Day 17 to healthy Japanese participants. Dose will be determined based on previous MRD cohorts.
  Interventions: Drug: TAK-988; Drug: TAK-988 Placebo

INTERVENTIONS:
Drug: TAK-988 — TAK-988 tablets.
Drug: TAK-988 Placebo — TAK-988 placebo-matching tablets.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of TAK-988 following single and multiple oral doses in healthy non-Japanese and Japanese adult participants and healthy elderly (HE) participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-988. TAK-988 is being tested to evaluate safety, tolerability, PK, and PD of single and multiple oral doses in healthy non-Japanese and Japanese adult participants and HE participants.

The study will enroll approximately 156 healthy participants. The study consists of 5 parts and up to 19 cohorts as mentioned below:

* TAK-988, Part A: Single-rising dose (SRD) design to assess the safety, tolerability, and PK of TAK-988 and effect of food on the PK of the TAK-988
* TAK-988, Part B: MRD design to assess the safety, tolerability, PK and PD of TAK-988
* TAK-988, Part C: MRD design to assess the safety, tolerability, PK and PD of TAK-988 and also central nervous system penetration relative to plasma concentrations of TAK-988
* TAK-988, Part D: MRD design to assess the safety, tolerability, PK and PD of TAK-988 for HE participants
* TAK-988, Part E: SRD and MRD design to assess the safety, tolerability, PK and PD of TAK-988 for Japanese origin participants

Participants in each cohort will be randomized to receive treatment with TAK-988 or matching placebo which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need).

This multi-center trial will be conducted in the United States. The overall duration of the study is approximately 10.5 months. Participants will make a final visit 7 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Be normotensive, with no history of hypertension or use of antihypertensive medication. Blood pressure (BP) must be less than (<) 140 millimeter of mercury (mmHg) (systolic) and <90 mmHg (diastolic).

   Healthy Adult and Elderly Participants (Parts A through D)
2. Must have a body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m^2) at the screening visit (non-Japanese only).

   Healthy Adult Participants (Parts A, B, and C)
3. Must be aged 18 to 55 years, inclusive, at the screening visit.
4. Must have a body weight >=50 kilogram (kg) at the screening visit.

   HE Participants (Part D)
5. Must be aged >=65 years, inclusive, at the time of informed consent.
6. Must have a body weight >=40 kg at the screening visit.

   Healthy Japanese Adult Participants (Part E)
7. Must be aged 18 to 55 years, inclusive, at the screening visit.
8. Must have a BMI >=18.0 and <=26.0 kg/m^2 at the screening visit.
9. Must have been born in Japan to a Japanese mother and father and have maternal and paternal Japanese grandparents.
10. Must have not been away from Japan for more than 10 years at the screening visit.
11. In the opinion of the investigator, must have a lifestyle that has not changed significantly since relocation from Japan.

Exclusion Criteria:

1. Has a known hypersensitivity to any component of the formulation of TAK-988 or related compounds.
2. Has a risk of suicide according to endorsement of Item 4 or 5 of the screening/baseline visit Columbia Suicide Severity Rating Scale (C-SSRS) or has made a suicide attempt in the previous 6 months.
3. Has a lifetime history of major psychiatric disorder, such as bipolar disorder or schizophrenia. Participant who have history of major depressive disorder (MDD) may be included, but participants who have current active MDD or who have had active MDD in the past 6 months are excluded.
4. Has a clinically significant history of head injury or head trauma.
5. Has a history of cerebral ischemia, transient ischemic attack, intracranial aneurysm, or arteriovenous malformation.
6. Screening electrocardiogram (ECG) reveals a QT interval with the Fridericia's correction method (QTcF) greater than (>) 450 millisecond (ms) (men) or >470 ms (women).
7. Has a resting heart rate outside of the range of 45 to 100 beats per minute, confirmed on repeat testing within a maximum of 30 minutes).

   Healthy Non-Japanese Adult Participants (Part C)
8. Has undergone CSF collection within 30 days before check-in (Day -2).
9. Has a known hypersensitivity to anesthesia or its derivatives used during CSF collection or to any medication used to prepare the area of lumbar puncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-17 (Estimated); Primary Completion 2022-04-29 (Estimated); Study Completion 2022-04-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) | Baseline up to Day 26
Number of Participants With at Least one Markedly Abnormal Value (MAV) for Laboratory Values | Baseline up to Day 26
Number of Participants With at Least one MAV for Vital Signs | Baseline up to Day 26
Number of Participants With at Least one MAV for Electrocardiograms (ECGs) | Baseline up to Day 26

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-988 | Day 1 (Parts A-E), Day 7 (Part C), Day 14 (Parts B and D), Day 17 (Part E) pre-dose and at multiple time points (up to 72 hours) post-dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-988 | Day 1 (Parts A-E), Day 7 (Part C), Day 14 (Parts B and D), Day 17 (Part E) pre-dose and at multiple time points (up to 72 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-988 | Day 1 (Parts A-E) pre-dose and at multiple time points (up to 72 hours) post-dose
AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-988 | Day 1 (Parts A-E) pre-dose and at multiple time points (up to 72 hours) post-dose
T1/2z: Terminal Disposition Phase Half-life for TAK-988 | Day 1 (Parts A-E) pre-dose and at multiple time points (up to 72 hours) post-dose
CLR: Renal Clearance for TAK-988 | Day 1 (Parts A, B, D and E), Day 14 (Parts B and D), Day 17 (Part E) pre-dose and at multiple time points (up to 72 hours) post-dose
AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to tau over Dosing Interval for TAK-988 | Day 7 (Part C), Day 14 (Parts B and D), Day 17 (Part E) pre-dose and at multiple time points (up to 72 hours) post-dose
Part C: Ratio of the Cerebrospinal Fluid (CSF) to Plasma AUC From Time 0 to 24 Hours for TAK-988 | Day 7 (Part C) Pre-dose and at multiple time points (up to 24 hours) post-dose
Rac (AUC): Accumulation Ratio Based on AUCτ for TAK-988 | Day 7 (Part C), Day 14 (Parts B and D), Day 17 (Part E) pre-dose and at multiple time points (up to 72 hours) post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Parexel Internalional - Glendale, Glendale, California
  - PRA Health Sciences - Salt Lake City, Millcreek, Utah

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.